CLINICAL TRIAL: NCT00686621
Title: Single Patient Emergency Treatment Use of Posaconazole in Invasive Fungal Infections
Brief Title: Single Patient Treatment of Posaconazole in Invasive Fungal Infections (Study P05113)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05113
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Posaconazole — Posaconazole oral suspension 400 mg twice daily with meal or nutritional supplement. Alternatively, if meal or nutritional supplement is not tolerated, posaconazole should be administered at a dose of 200 mg four times a day.
  Other Names: SCH 056592

SUMMARY:
The purpose of this study is to provide posaconazole compassionate treatment to patients with invasive fungal infections: 1) which are resistant to standard antifungal therapies; 2) for which there are no effective therapies; 3) with a prior history of serious, severe, or life-threatening toxicities while receiving standard antifungal therapies, or 4) with pre-existing organ dysfunction which precludes the use of standard antifungal therapies.

DETAILED DESCRIPTION:
NCT00686621 was voluntarily registered even though it is a single patient use study, also known as compassionate exemption study; therefore results will not be disclosed for this study.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Adults (age >=18 years) of either gender and of any race.
* Children (age >= 2 to 17 years) of either gender and of any race, who are not eligible for enrollment under any current clinical trial. Compassionate use will be permitted only under the direct supervision of qualified experts in pediatric infectious diseases with the written approval of the Schering Plough medical director (local country operations or headquarters project director).
* Subject or his/her legally authorized representative has given signed, written informed consent,
* Ability to take study medication orally by swallowing or via an enteral feeding tube.
* Subject is not considered eligible for any other clinical research program with posaconazole.

Safety Related Inclusion Criteria

* Male or a female patient who meets any one of the following criteria:

  * postmenopausal, surgically sterilized, or documented to have primary ovarian failure due to prior cytotoxic chemotherapy or radiation therapy; abstinent from sexual intercourse or practicing effective birth control. Effective birth control methods must continue for at least 30 days after discontinuation of treatment with posaconazole.
* Known to be non pregnant by history or (preferably) by negative serum or urine pregnancy test prior to the first dose of posaconazole for all females of childbearing potential.
* Not breast feeding or if lactating, willing to discontinue breast feeding during treatment.

Invasive Fungal Infection Inclusion Criteria

* Each patient must have:

  * A documented invasive fungal infection who have failed a reasonable trial of other licensed antifungal agents, either due to progression or lack of improvement of the infection, or
  * Serious, severe or life-threatening toxicities related to current or prior antifungal therapy, or
  * An invasive fungal infection for which there are currently no effective therapies.
* Patients with debilitating but not immediately life threatening fungal diseases, where significant morbidity may result in disability and where prior antifungal therapy has been unsuccessful (eg, chronic mucocutaneous candidiasis, recurrent oropharyngeal or esophageal candidiasis with dehydration and malnutrition, or cutaneous phaeohyphomycosis and mycetoma).

Exclusion Criteria:

* Women who are pregnant or who will continue to breast-feed infants.
* History of serious or severe hypersensitivity or idiosyncratic reactions to azole antifungals.
* Patients who require ongoing treatment with any prohibited medication (see Core Clinical Data Sheet and list of Prohibited Medications) and for whom an appropriate washout period has not elapsed.
* Patients who are in a situation or have any condition requiring the use of prohibited drugs or unstable medical conditions where the risk of therapy would exceed any potential benefit i.e., hematological disorder such as unstable cardiac disorder (including acute myocardial infarction or unstable myocardial ischemia/angina within 30 days, ventricular arrhythmia within 30 days, uncontrolled atrial fibrillation, or atrial fibrillation/flutter with symptomatic bradycardia [sick sinus syndrome], or unstable congestive heart failure) or impairment expected to be unstable or progressive during the course of this study (e.g., recurrent or uncontrolled seizure disorders, demyelinating syndromes, or progressive peripheral neuropathy).
* Patients receiving vinca alkaloids or anthracyclines within 24 hours of study enrollment or requiring therapy with vinca alkaloids or anthracyclines within the next 30 days for treatment of uncontrolled (pre-existing) malignancy or requiring ongoing therapy with vinca alkaloids or anthracyclines, where the risk of toxicity from these medicinal products is considered to be significant.
* Any condition requiring the use of prohibited drugs (please consult current product labeling).
* Hepatic function tests: alanine amino transferase (ALT) or aspartate aminotransferase (AST) >10 times upper limit of normal, or evidence of severe hepatic dysfunction based on other clinical assessment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult